#### ASSENT TO BE IN A RESEARCH STUDY

# Remote School-Home Program to Improve Youth Attention and Behavior in Mexican Students For children 7 – 12 years old

## Why are we meeting with you?

We want to tell you about something we are doing called a research study. A research study is when doctors collect a lot of information to learn more about something. Dr. Eva Araujo and some other doctors are doing a study to learn more about how to help children make friends and do better in school. After we tell you about it, we will ask if you'd like to be in this study or not.

### Why are we doing this study?

We are doing a study that looks at ways to help children. We are hoping to learn more about the kinds of things that might help children do better at school and get along better with other kids and their families. In the whole study, there will be about 88 kids and their families.

## What will happen to you if you are in the study?

If you agree to be in the study, this is what will happen:

We will ask you and your parents and teachers questions about how you are doing at home, at school and with friends.

Then, either very soon or spring of this school year, which is decided by chance(like flipping a coin), you will be in a remote group with other children at your school over videoconferencing. This group will meet 6 times for about one hour each time. You will learn new ways to get along with others, play games, and stay organized. The group is meant to be fun. You will also meet with your group leader and your parents and teacher one time for about half an hour to go over things you learned in the group.

#### Will any parts of the study hurt?

Nothing in the study will hurt you. You may feel uncomfortable about answering some of the questions, but your answers may help us learn about how children get along with their parents and with other children. You may skip any questions you do not want to answer.

## Will you get better if you are in this study?

We don't know for sure. You might not get any better. Or, you might do better in school or you might get along better with friends and family.

## Do you have any questions?

You can ask questions any time. You can ask now. You can ask later. You can talk to me or you can talk to someone else.

## Do you have to be in this study?

No, you don't. No one will be mad at you if you don't want to do this. If you don't want to be in this study, just tell us. Or if you do want to be in the study, tell us that. And, remember, you can say yes now and change your mind later. It's up to you.

Assent Form

If you don't want to be in this study, just say so. If you want to be in this study, please tell me "Yes, I want to be in the study."

| Your family will be given a copy of this form to keep. | |
|---|---|
| SIGNATURE OF PERSON CONDUCTING ASSENT DISC | CUSSION |
| I have explained the study tounderstand, and the child has verbally agreed to be in the study. | (child name) in language he/she can |
| Signature of Person Conducting Assent Discussion | Date |
| Name of Person Conducting Assent Discussion (print) | |